CLINICAL TRIAL: NCT06918158
Title: Comparative Study on the Effectiveness of Mobilization With Movement Versus Joint Specific Manipulation on Pain and Function in Patient With Dequervains Tenosynovitis
Brief Title: Mobilization With Movement Versus Joint-Specific Manipulation in De Quervain's Tenosynovitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC-01001 Khaista Bacha
Record Dates: First submitted 2025-02-20; First posted 2025-04-09 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Tenosynovitis
Keywords: Tenosynovitis
MeSH Terms: conditions — Tenosynovitis | interventions — Movement

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Joint-specific Manipulation (Experimental): Group A
  Interventions: Other: Joint Specific Manipulation
- Mobilization with Movement (Placebo Comparator): Group B
  Interventions: Other: Mobilization with Movement

INTERVENTIONS:
Other: Mobilization with Movement — Mobilization with Movement
  * The proximal row of carpals glides passively radially.
  * Active thumb and wrist movements superimposed on the glide.
  Therapeutic excercises:
  * Ball Toss
  * Static web gripping
  * Gentle ROM activities to maintain mobility
  * Isometric exercises in all direction
  Arms: Mobilization with Movement
Other: Joint Specific Manipulation — Joint Specific Manipulation
  * High-velocity, low-amplitude thrust to the first carpometacarpal joint
  * Radiocarpal wrist mobilization .Grade III-IV applied at end range. 2. Therapeutic excercises:
  * Ball Toss
  * Static web gripping
  * Gentle ROM activities to maintain mobility
  * Isometric exercises in all direction Ergonomics modifications
  Arms: Joint-specific Manipulation

SUMMARY:
A comparative study on the effectiveness of mobilization with movement (MWM) versus joint-specific manipulation (JSM) in patients with De Quervain's tenosynovitis typically aims to assess how each technique impacts pain relief and functional improvement. De Quervain's tenosynovitis is an inflammation of the tendons around the thumb and wrist, often causing pain, swelling, and difficulty in performing everyday tasks. The study would likely compare the two interventions by measuring pain levels, range of motion, and overall functional outcomes before and after treatment. MWM involves applying specific, controlled movements while the patient is actively engaging in their joint motion, targeting the tissue's mobility and reducing pain. JSM, on the other hand, focuses on manipulating the joint directly to restore normal function, specifically targeting the wrist and thumb regions affected by the condition.

DETAILED DESCRIPTION:
A comparative study on the effectiveness of Mobilization with Movement (MWM) versus Joint-Specific Manipulation (JSM) in patients with De Quervain's Tenosynovitis would delve deeper into the physiological mechanisms and clinical outcomes associated with each technique, providing valuable evidence for therapeutic decision-making. De Quervain's Tenosynovitis is a condition characterized by the inflammation of the tendons at the base of the thumb, particularly affecting the abductor pollicis longus and extensor pollicis brevis tendons. This condition is commonly caused by repetitive strain, overuse, or trauma, leading to pain, swelling, and restricted movement, which significantly impacts the patient's daily activities.

ELIGIBILITY:
Inclusion Criteria:o Patients clinically diagnosed with De Quervain's tenosynovitis

* Age between 25-45 years.
* Positive Finkelstein test.
* Pain over the first dorsal compartment.
* Limited wrist and thumb function.
* Willingness to take part and adhere to the study's guidelines.

Exclusion Criteria:Participants fall in this category would be excluded of the study.

* Previous surgery of wrist or thumb.
* Presence of neurological symptoms like numbness, weakeness.
* Rheumatological conditions like rheumatoid arthritis.
* Pregnancy.
* Presence of wrist fracture or osteoporosis.
* Carpel tunnel syndrome.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Pain Reduction - Measured using the Numeric Pain Rating Scale (NPRS) (0-10 scale). | 6 Months
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS), a validated tool where participants rate their pain on a scale from 0 no pain to 10 worst possible pain.

SECONDARY OUTCOMES:
Wrist Function - Assessed with the Patient-Rated Wrist Evaluation (PRWE) (0-100 scale). | 6months
  Functional wrist use will be assessed using the Patient-Rated Wrist Evaluation (PRWE), which evaluates pain and disability on a 100-point scale, with higher scores indicating greater impairment. Clinical signs will be assessed using Finkelstein's Test, a standard diagnostic test for De Quervain's tenosynovitis, recorded as positive or negative. Data will be analyzed using pre- and post-intervention comparisons within and between groups to determine the effectiveness of each intervention.

OTHER OUTCOMES:
Clinical Signs - Evaluated using Finkelstein's Test (Positive/Negative). | 6 months
  Clinical Signs will be assessed using Finkelstein's Test, recorded as positive or negative based on the presence of pain during the maneuver.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Nadeem Ahmad, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University Malakand Campus, Malakand, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No